CLINICAL TRIAL: NCT02214147
Title: Pharmacokinetics of Oral Alisertib (MLN8237) in Adult Patients With Advanced Solid Tumors or Relapsed/Refractory Lymphoma With Varying Degrees of Hepatic Function
Brief Title: Pharmacokinetics of Alisertib in Adults With Advanced Solid Tumors or Relapsed/Refractory Lymphoma With Varying Degrees of Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C14019; U1111-1155-6072 (Other: World Health Organization)
Record Dates: First submitted 2014-07-30; First posted 2014-08-12 (Estimated); Results first posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-04

CONDITIONS: Advanced Solid Tumors; Relapsed/Refractory Lymphoma
Keywords: Drug Therapy
MeSH Terms: conditions — Lymphoma | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alisertib: Normal Hepatic Function (Experimental): Alisertib 50 mg, orally, once, on Cycle 1 Day 1, followed by, alisertib 50 mg, orally, twice daily (BID) for 7 days (Cycle 1 Day 8 to 14) followed by a 14-day rest period. Starting at Cycle 2 Day 1, alisertib 50 mg, BID for 7 days, followed by a 14-day rest period unless a dose reduction is indicated. Participants may continue to receive alisertib until they experience progressive disease or unacceptable alisertib-related toxicities for up to 12 months (approximately 16 cycles), unless it is determined by the investigator, with agreement by the sponsor, that a participant would derive clinical benefit from continued treatment beyond 12 months. Normal hepatic function includes participants with total bilirubin ≤ upper limit of the normal range [ULN] and alanine aminotransferase [ALT] level ≤ ULN.
  Interventions: Drug: Alisertib
- Alisertib: Moderate Hepatic Impairment (Experimental): Alisertib 50 mg, orally, once, on Cycle 1 Day 1, followed by alisertib 30 mg, BID for 7 days (Cycle 1 Day 8 to 14), followed by a 14-day rest period. Starting at Cycle 2 Day 1, alisertib 30 mg, BID for 7 days followed by a 14-day rest period unless a dose reduction is indicated. Participants may continue to receive alisertib until they experience progressive disease or unacceptable alisertib-related toxicities for up to 12 months (approximately 16 cycles), unless it is determined by the investigator, with agreement by the sponsor, that a participant would derive clinical benefit from continued treatment beyond 12 months. Moderate hepatic impairment includes participants with total bilirubin > 1.5-3 x ULN and any ALT level.
  Interventions: Drug: Alisertib
- Alisertib: Severe Hepatic Impairment (Experimental): Alisertib 50 mg, orally, once, on Cycle 1 Day 1, followed by, alisertib 20 mg, BID for 7 days (Cycle 1 Day 8 to 14) followed by a 14-day rest period. Starting at Cycle 2 Day 1, alisertib 20 mg, BID for 7 days followed by a 14-day rest period unless a dose reduction is indicated. Participants may continue to receive alisertib until they experience progressive disease or unacceptable alisertib-related toxicities for up to 12 months (approximately 16 cycles), unless it is determined by the investigator, with agreement by the sponsor, that a participant would derive clinical benefit from continued treatment beyond 12 months. Severe hepatic impairment includes participants with total bilirubin > 3 x ULN and any ALT level.
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — Alisertib will be supplied as enteric coated tablets.
  Other Names: MLN8237

SUMMARY:
The purpose of this study is to evaluate the effect of moderate or severe hepatic impairment on the single-dose pharmacokinetics of alisertib in adult participants with cancer.

DETAILED DESCRIPTION:
The drug being tested in this study is called alisertib. Alisertib was tested to assess how it was processed by the body in participants with advanced solid tumors or relapsed/refractory lymphoma with varying degrees of liver function. This study also assessed laboratory results and safety.

The study enrolled 36 participants. Participants were assigned to 1 of the 3 treatment groups based on the status of their liver function: Normal hepatic function (Total bilirubin ≤ upper limit of the normal range [ULN] and alanine aminotransferase [ALT] level ≤ ULN), moderate hepatic impairment (Total bilirubin > 1.5-3 x ULN and ALT level = Any), or severe hepatic impairment (Total bilirubin > 3 x ULN and ALT level = Any). All participants were administered one 50 mg dose of alisertib on Day 1, Cycle 1. Alisertib was administered again on Days 8 through 14 of Cycle 1, followed by a 14-day rest period. Doses administered on Days 8-14 were 50, 30, or 20 mg of alisertib, depending on hepatic function. Alisertib was then continued at the same dose as in Cycle 1, Days 8-14 in 21-day cycles (7 days of alisertib followed by a 14-day rest period) for up to 1 year (approximately 16 cycles).

This multicenter trial was conducted in USA only. The overall time to participate in this study was up to 312 Days. Participants made multiple visits to the clinic including an end-of-study visit 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants 18 years of age or older.
2. Histologically or cytologically confirmed metastatic and/or advanced solid tumors or lymphomas for which standard curative or life-prolonging treatment does not exist or is no longer effective or tolerable.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
4. Female participants who:

   * Are post-menopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study drug, or agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant (periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception).
5. Male participants, even if surgically sterilized (ie, status postvasectomy), who:

   * Agree to practice effective barrier contraception during the entire study treatment period and through 4 months after the last dose of study drug, or
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant (periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception).
6. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
7. Suitable venous access for the study-required blood sampling, including pharmacokinetics.
8. Ability to swallow tablets.
9. Participants with biliary obstruction for which a stent had been placed are eligible provided that the stent has been in place for more than 14 days before the first dose of alisertib and liver function has stabilized.
10. Recovered from the reversible effects of prior antineoplastic therapy (ie, ≤ Grade 1 toxicity or baseline).
11. Clinical laboratory values as specified below:

    * Absolute neutrophil count (ANC) ≥ 1500/μL and platelet count ≥ 75,000/μL.

      * Participants with normal hepatic function: Total bilirubin and alanine aminotransferase (ALT) must be ≤ upper limit of the normal range (ULN).
      * Participants with moderate hepatic impairment: total bilirubin must be > 1.5 to 3 x ULN with any ALT level.
      * Participants with severe hepatic impairment: total bilirubin must be > 3 x ULN with any ALT level.
      * Measured creatinine clearance or calculated creatinine clearance > 30 mL/minute. Note: If a calculated creatinine clearance is used, it should be calculated according to the Cockcroft-Gault formula.
      * Hemoglobin must be ≥ 8 g/dL.

Exclusion Criteria:

1. Participants of North/East Asian ethnicity (ie, Japanese, Chinese, Korean) will be excluded.
2. Recurrent nausea and/or vomiting within 14 days before the first dose of alisertib or known gastrointestinal (GI) abnormality or GI procedure that could interfere with or modify the oral absorption or tolerance of alisertib. Examples include, but are not limited to, disease-related bowel obstruction, pancreatic insufficiency, use of pancreatic enzymes, a gastric condition (such as severe reflux or active peptic ulcer disease) that requires chronic and uninterrupted use of proton pump inhibitors, partial gastrectomy, history of small intestine surgery, and celiac disease.
3. Participants requiring treatment with clinically significant enzyme inducers, such as the enzyme-inducing anti-epileptic drugs phenytoin, carbamazepine, phenobarbital, oxcarbazepine, primidone, rifampin, rifabutin, rifapentine, or St. John's wort within 14 days before the first dose of alisertib or requiring the use of these medications during the study.
4. A medical condition requiring use of pancreatic enzymes; daily, chronic, or regular use of proton pump inhibitors (PPIs); or histamine 2 (H2) receptor antagonists. Participants who intermittently use these medications, must meet the following criteria:

   * No use of PPIs within 5 days before the first dose of alisertib.
   * No use of H2 antagonist or pancreatic enzymes within 24 hours before the first dose of alisertib.
5. Inadequate bone marrow or other organ function (excluding hepatic impairment per eligibility criteria).
6. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period or a positive urine pregnancy test on Day 1 before first dose of alisertib.
7. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
8. Treatment with any anticancer therapy or any investigational products within 3 weeks before the first dose of study drug.
9. Exposure to nitrosoureas or mitomycin C within 42 days before the first dose of study drug.
10. Radiotherapy within 14 days before the first dose of study drug.
11. Prior treatment with radiation therapy involving ≥ 25% of the hematopoietically active bone marrow within 42 days before the first dose of study drug.
12. Major surgery within 14 days before the first dose of study drug.
13. Serious infection within 14 days before the first dose of study drug. Participant must have recovered from infection before first dose.
14. Life-threatening illness unrelated to cancer.
15. Symptomatic brain metastasis. Participants with brain metastases:

    * Must have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks after completion of the definitive therapy AND
    * Must be without neurologic dysfunction that would confound the evaluation of neurologic or other adverse events (AEs).
16. Clinically significant coagulopathy or bleeding disorder.
17. Severe central nervous system, pulmonary, or renal disease not related to the participant's cancer.
18. Known human immunodeficiency virus (HIV) positive.
19. Known history of hepatitis C infection or suspected currently active hepatitis C infection, or known or suspected history of hepatitis B infection. Participants with known or suspected history of hepatitis B infection were to be screened and excluded when any of the following conditions were met:

    * Received hematopoietic stem cell transplantation (either allogeneic or autologous), or
    * Received any rituximab-containing treatment regimen in the last 12 months before entering the study, or
    * Tested positive for the presence of at least 1 of the following 3 markers in blood (evaluated at Screening): hepatitis B surface antigen (HBsAg), antibodies against hepatitis B core antigen (anti-HBc), or hepatitis B virus deoxyribonucleic acid (HBV DNA).
20. Any of the following cardiovascular conditions:

    * Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
    * Corrected QT interval (QTc) > 500 milliseconds in a 12-lead electrocardiogram (ECG) during screening.
21. History of uncontrolled sleep apnea syndrome or other condition that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease.
22. Use of moderate or strong cytochrome P450 (CYP) 3A inhibitors or CYP3A inducers within 2 weeks before the first dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-08-21 (Actual); Primary Completion 2016-04-05 (Actual); Study Completion 2016-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (7):
- United States (7):
  - Miami, Florida
  - Chicago, Illinois
  - Ann Arbor, Michigan
  - St Louis, Missouri
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 6 investigative sites in the United States from 21 August 2014 to 18 July 2016.
Pre-assignment Details: Participants with a diagnosis of advanced solid tumors or relapsed/refractory lymphoma were assigned to 1 of 3 hepatic function groups (normal hepatic function, moderate hepatic impairment, or severe hepatic impairment) on the basis of their total bilirubin and alanine aminotransferase (ALT) values. All participants received alisertib.
Period: Overall Study
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Started | 16 | 12 | 8
Completed (Completed=Completed protocol-specified dosing and PK assessment.) | 16 | 12 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population was defined as all participants who received at least 1 dose of alisertib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment | Total
Number analyzed (Participants) | 16 | 12 | 8 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.07) | 54.9 (9.89) | 54.0 (7.05) | 57.5 (9.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 2 | 14
  Male | 11 | 5 | 6 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 14 | 11 | 6 | 31
  Not Reported | 1 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 14 | 11 | 6 | 31
  Black or African American | 2 | 1 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16 | 12 | 8 | 36
Height [Mean (Standard Deviation); unit: cm] — Population: Height data is only available for n=14,11,5 participants.
  cm
    number analyzed (Participants) | 14 | 11 | 5 | 30
    (all) | 172.9 (14.62) | 162.9 (7.79) | 178.2 (8.10) | 170.1 (12.66)
Weight [Mean (Standard Deviation); unit: kg] | 84.6 (20.997) | 85.5 (33.881) | 85.8 (11.847) | 85.2 (24.044)
Body surface area [Mean (Standard Deviation); unit: m^2] — Body surface area=square root[height(cm)*weight(kg)/3600] Population: Body surface area data is only available for n=14,11,5 participants.
  m^2
    number analyzed (Participants) | 14 | 11 | 5 | 30
    (all) | 2.030 (0.3073) | 1.897 (0.4028) | 2.056 (0.1970) | 1.986 (0.3292)

OUTCOME MEASURES:

1. Primary Outcome: Unbound Cmax: Maximum Observed Plasma Concentration for Alisertib
Time Frame: Cycle 1 Day 1 Pre-dose and, and at multiple timepoints (up to 168 hours) post-dose
Population: Pharmacokinetic (PK)-evaluable population was defined as all participants who had completed protocol-specified dosing and PK assessment in Cycle 1 with sufficient dosing and PK data to reliably estimate PK parameters.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Number analyzed (Participants) | 16 | 12 | 8
nmol/L | 17.3 (9.09) | 28.1 (7.82) | 18.5 (5.80)
Statistical Analysis 1: Comparison: Alisertib: Normal Hepatic Function vs Alisertib: Moderate Hepatic Impairment vs Alisertib: Severe Hepatic Impairment; Test type: Other — The effect of hepatic impairment on alisertib PK. Combined analysis of moderate and severe hepatic impairment in reference to normal hepatic function; Least Squares Geometric Mean Ratio = 1.42, 90% CI 2-sided [1.12 to 1.80] — Least Squares Geometric Means Ratio= Moderate + Severe Hepatic Impairment/Normal Hepatic Function

2. Primary Outcome: Unbound AUClast: Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Alisertib
Time Frame: Cycle 1 Day 1 Pre-dose and, and at multiple timepoints (up to 168 hours) post-dose
Population: Participants from the PK-evaluable population, all participants who had completed protocol-specified dosing and PK assessment in Cycle 1 with sufficient dosing and PK data to reliably estimate PK parameters, with data available for analysis.
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Number analyzed (Participants) | 16 | 10 | 8
h*nmol/L | 248.5 (131.41) | 859.1 (387.85) | 735.4 (444.61)
Statistical Analysis 1: Comparison: Alisertib: Normal Hepatic Function vs Alisertib: Moderate Hepatic Impairment vs Alisertib: Severe Hepatic Impairment; Test type: Other — [test comment as in outcome 1, analysis 1]; Least Squares Geometric Mean Ratio = 3.21, 90% CI 2-sided [2.33 to 4.43] — Least Squares Geometric Mean Ratio=Moderate + Severe Hepatic Impairment/Normal Hepatic Function

3. Primary Outcome: Unbound AUC0-∞: Area Under the Concentration-Time Curve From Time 0 to Infinity for Alisertib
Time Frame: Cycle 1 Day 1 Pre-dose and, and at multiple timepoints (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Number analyzed (Participants) | 12 | 10 | 7
h*nmol/L | 304.3 (119.09) | 937.6 (428.98) | 778.0 (610.51)
Statistical Analysis 1: Comparison: Alisertib: Normal Hepatic Function vs Alisertib: Moderate Hepatic Impairment vs Alisertib: Severe Hepatic Impairment; Test type: Other — [test comment as in outcome 1, analysis 1]; Least Squares Geometric Mean Ratio = 2.54, 90% CI 2-sided [1.84 to 3.53] — Least Squares Geometric Mean Ratio=Moderate + Severe Hepatic Impairment/Normal Hepatic Function

4. Secondary Outcome: Percentage of Participants Who Experienced at Least 1 Treatment-Emergent Adverse Event
Description: An adverse event is any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline to 30 days after last dose (Up to 312 Days)
Population: Safety population was defined as all participants who received at least 1 dose of alisertib.
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Number analyzed (Participants) | 16 | 12 | 8
percentage of participants | 100 | 100 | 100

5. Secondary Outcome: Percentage of Participants Who Experienced at Least 1 Serious Adverse Event
Description: A serious adverse event is any untoward medical occurrence or effect that at any dose of a drug results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is medically important due to other reasons than the above mentioned criteria.
Time Frame: Baseline to 30 days after last dose (Up to 312 Days)
Population: Safety population was defined as all participants who received at least 1 dose of alisertib.
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Number analyzed (Participants) | 16 | 12 | 8
percentage of participants | 44 | 67 | 88

6. Secondary Outcome: Percentage of Participants With Clinically Significant Laboratory Values
Description: Laboratory assessments include serum chemistry and hematology. An abnormal laboratory value was assessed as an AE if that value led to discontinuation or delay in treatment, dose modification, therapeutic intervention, or was considered by the investigator to be a clinically significant change from baseline.
Time Frame: Baseline to the end of the study (Up to 312 Days)
Population: Safety population was defined as all participants who received at least 1 dose of alisertib.
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Number analyzed (Participants) | 16 | 12 | 8
percentage of participants
  Gamma-glutamyltransferase increased | 13 | 0 | 0
  Alanine aminotransferase increased | 0 | 8 | 0
  Aspartate aminotransferase increased | 0 | 8 | 0
  Blood bilirubin increased | 0 | 8 | 0
  Transaminases increased | 0 | 8 | 0
  Blood sodium decreased | 6 | 8 | 0
  Blood calcium increased | 6 | 0 | 0
  Blood phosphorus decreased | 6 | 0 | 0
  Platelet count decreased | 6 | 8 | 0
  Blood alkaline phosphatase increased | 6 | 8 | 0
  Blood creatinine increased | 0 | 8 | 0
  Neutrophil count decreased | 0 | 8 | 0
  White blood cell count decreased | 0 | 8 | 0

7. Secondary Outcome: Percentage of Participants With Clinically Significant Vital Signs
Description: Vital signs include measurements of sitting diastolic and systolic blood pressure, heart rate, and temperature. Any vital signs determined by the investigator to be clinically significant were recorded as AEs.
Time Frame: Baseline to the end of the study (Up to 312 days)
Population: Safety population was defined as all participants who received at least 1 dose of alisertib.
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Number analyzed (Participants) | 16 | 12 | 8
percentage of participants
  Pyrexia | 25 | 8 | 38
  Sinus tachycardia | 6 | 0 | 0

8. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Alisertib Metabolites M1 and M2
Time Frame: Cycle 1 Day 1 Pre-dose and, and at multiple timepoints (up to 168 hours) post-dose
Population: PK-evaluable population was defined as all participants who had completed protocol-specified dosing and PK assessment in Cycle 1 with sufficient dosing and PK data to reliably estimate PK parameters.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Number analyzed (Participants) | 16 | 12 | 8
nmol/L
  Metabolite M1 | 370.3 (282.02) | 1774.0 (904.10) | 2001.9 (1094.75)
  Metabolite M2 | 154.6 (82.54) | 173.8 (54.39) | 207.3 (151.60)

9. Secondary Outcome: Tmax: Time of First Occurrence of Cmax for Alisertib Metabolites M1 and M2
Time Frame: Cycle 1 Day 1 Pre-dose and, and at multiple timepoints (up to 168 hours) post-dose
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Number analyzed (Participants) | 16 | 12 | 8
hours
  Metabolite M1 | 3.500 [1.88 to 7.92] | 24.000 [1.00 to 48.30] | 24.150 [9.08 to 96.70]
  Metabolite M2 | 9.000 [5.88 to 49.30] | 24.050 [9.00 to 72.10] | 24.150 [9.08 to 96.70]

10. Secondary Outcome: AUClast: Area Under the Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Alisertib Metabolites M1 and M2
Description: The area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUC0-last) of the alisertib metabolites M1 and M2 was determined from the concentration-time curve of each participant using non-compartmental methods.
Time Frame: Cycle 1 Day 1 Pre-dose and, and at multiple timepoints (up to 168 hours) post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Number analyzed (Participants) | 16 | 10 | 8
h*nmol/L
  Metabolite M1 | 8366.3 (10790.88) | 159665.0 (116960.23) | 196750.0 (117472.08)
  Metabolite M2 | 8923.1 (6539.00) | 17326.0 (8562.96) | 16987.5 (9384.25)

11. Secondary Outcome: Dose-normalized Trough Concentration of Alisertib on Cycle 1 Day 14
Description: A single blood sample will be collected pre-dose on Cycle 1 Day 14. The concentration of alisertib was determined in the plasma sample and dose-normalized.
Time Frame: Pre-dose on Day 14 of Cycle 1
Population: Data was not collected, as many participants dropped out of the study prior to Day 14 trough concentration collection.
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose of study drug to 30 days past last dose (Up to 312 Days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alisertib: Normal Hepatic Function | Alisertib: Moderate Hepatic Impairment | Alisertib: Severe Hepatic Impairment
All-Cause Mortality (participants affected / at risk) | 2/16 | 3/12 | 4/8
Serious Adverse Events (participants affected / at risk) | 7/16 | 8/12 | 7/8
Other Adverse Events (participants affected / at risk) | 15/16 | 12/12 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib: Normal Hepatic Function (N=16) | Alisertib: Moderate Hepatic Impairment (N=12) | Alisertib: Severe Hepatic Impairment (N=8)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Pancreatic neuroendocrine tumour metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 0 | 1
Malaise (General disorders) | 1 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 — One treatment-emergent death occurred during treatment with alisertib and is not related.
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib: Normal Hepatic Function (N=16) | Alisertib: Moderate Hepatic Impairment (N=12) | Alisertib: Severe Hepatic Impairment (N=8)
Nausea (Gastrointestinal disorders) | 9 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 6 | 4 | 0
Vomiting (Gastrointestinal disorders) | 4 | 4 | 0
Ascites (Gastrointestinal disorders) | 0 | 6 | 1
Constipation (Gastrointestinal disorders) | 5 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 0 | 0
Retching (Gastrointestinal disorders) | 1 | 2 | 0
Gingival pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Eructation (Gastrointestinal disorders) | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 1 | 0 | 0
Fatigue (General disorders) | 6 | 3 | 3
Pyrexia (General disorders) | 4 | 1 | 2
Oedema peripheral (General disorders) | 2 | 3 | 1
Chills (General disorders) | 4 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0
Mass (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 3 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 5 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 3 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 1 | 1
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 | 1 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Tongue biting (Nervous system disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 3 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 3 | 2
Anxiety (Psychiatric disorders) | 1 | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Stress (Psychiatric disorders) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0
Blood sodium decreased (Investigations) | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Blood calcium increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 5 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 2 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1
Eye irritation (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.